CLINICAL TRIAL: NCT00304135
Title: Randomized Phase II-III Study of Chemoradiation With Fluorouracil and Cisplatin Versus Chemotherapy (Gemcitabine/Oxaliplatin) in Non Resectable But Non Metastatic Cancer of the Biliary Tract
Brief Title: Fluorouracil, Cisplatin, and Radiation Therapy or Gemcitabine and Oxaliplatin in Treating Patients With Nonmetastatic Biliary Tract Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000470411; FFCD-9902; SANOFI-FFCD-9902; LILLY-FFCD-9902; FFCD-FNCLCC-SFRO-9902
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2006-12

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: localized unresectable adult primary liver cancer; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms | interventions — Cisplatin; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radio-chimiothérapie (Active Comparator): Radio-chimiothérapie
  Interventions: Drug: cisplatin
- GEMOX (Experimental): GEMOX
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: cisplatin
  Arms: Radio-chimiothérapie
Drug: gemcitabine hydrochloride
  Arms: GEMOX
Drug: oxaliplatin
  Arms: GEMOX

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, cisplatin, oxaliplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether giving fluorouracil and cisplatin together with radiation therapy is more effective than giving gemcitabine together with oxaliplatin in treating nonmetastatic biliary tract cancer.

PURPOSE: This randomized phase II/III trial is studying fluorouracil, cisplatin, and radiation therapy to see how well they work compared to gemcitabine and oxaliplatin in treating patients with nonmetastatic biliary tract cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the 3-month progression rate in patients with unresectable, nonmetastatic cancer of the biliary tract treated with fluorouracil, cisplatin, and radiotherapy vs gemcitabine hydrochloride and oxaliplatin. (phase II)
* Compare the overall survival of patients treated with these regimens. (phase III)

Secondary

* Compare toxicities of these regimens in these patients. (phase II)
* Compare the quality of life at initial drainage (phase II) and overall (phase III) of patients treated with these regimens.
* Compare the biliary complication rate in patients treated with these regimens.
* Compare the duration of hospitalization of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease location (gallbladder vs intrahepatic biliary duct vs extrahepatic biliary duct). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily, 5 days a week on days 1-33. Patients also receive fluorouracil IV continuously over 5 days once a week in weeks 1-5 and cisplatin IV over 15 minutes on days 1-4 and 29-32 (or days 1 or 2 and 29 or 30) in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine hydrochloride IV over 100 minutes and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 3 months thereafter.

After completion of study therapy, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 170 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer of the biliary tract by 1 of the following methods:

  * Histologic confirmation
  * Stenosis of the biliary tract by MRI, CT scan, or ECHO
* Unresectable disease
* Amenable to radiotherapy
* No visceral metastases by imaging

  * Hepatic adenopathies that can be included in a radiation field allowed
* No known ampulla of Vater or pancreatic cancer involving the biliary tract

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Creatinine < 1.5 mg/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Prothrombin time > 70%
* Bilirubin ≤ 2.9 mg/dL (after hepatic draining, if needed)
* No unstable angina
* No symptomatic cardiac insufficiency
* No other comorbidity that would preclude study therapy
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No prior hydatid cyst or alveolar echinococciasis
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No recent biliary surgery
* No hepatic intra-arterial chemotherapy
* No prior anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression rate at 3 months | 2012
Overall survival | 2012

SECONDARY OUTCOMES:
Toxicity | 2012
Biliary complication rate | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Chauffert, Principal Investigator — Centre Georges Francois Leclerc
Locations (20):
- France (20):
  - Centre Hospitalier General, Belfort
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier de Dax, Dax
  - Hopital Du Bocage, Dijon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - C. H. Du Mans, Le Mans
  - CHU de la Timone, Marseille
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Bichat - Claude Bernard, Paris
  - CHU Pitie-Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Sebastopol, C.H.U. de Reims, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Hospitalier de Semur en Auxois, Semur-en-Auxois
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier de Tarbes, Tarbes

REFERENCES:
- [Result] Phelip JM, Vendrely V, Rostain F, Subtil F, Jouve JL, Gasmi M, Michel P, Le Malicot K, Smith D, Seitz JF, Fauchart JP, Martin P, Bennouna J, Morin T, Bonnet I, Maingon P, Lepage C, Chauffert B. Gemcitabine plus cisplatin versus chemoradiotherapy in locally advanced biliary tract cancer: Federation Francophone de Cancerologie Digestive 9902 phase II randomised study. Eur J Cancer. 2014 Nov;50(17):2975-82. doi: 10.1016/j.ejca.2014.08.013. Epub 2014 Sep 17. PMID 25241229